CLINICAL TRIAL: NCT03463343
Title: Neurophysiologic Effects of Cervical Spinal Manipulation in Asymptomatic Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Escola Superior de Tecnologia da Saúde do Porto (Other)
Responsible Party: Principal Investigator, Nuno Filipe Pinho Nogueira, Invited Professor, Escola Superior de Tecnologia da Saúde do Porto
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20122017
Record Dates: First submitted 2017-09-08; First posted 2018-03-13 (Actual); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Manual manipulation (Experimental): In the Manual manipulation group, the thrust was applied in the right side of C3/C4 with neutral flexion/extension, ipsilateral side bending and contralateral rotation. Then, a low amplitude, high velocity thrust in rotation was delivered.
  Interventions: Other: Cervical spine manual manipulation
- Mechanical manipulation (Active Comparator): In the Mechanical manipulation group, the Activator instrument was applied on the right transverse apophyses of C3.
  Interventions: Other: Cervical spine mechanical manipulation
- Placebo (Placebo Comparator): The subjects were positioned in the same pre-manipulative position as the manual manipulation group, but the thrust didn't occur. Instead, the position was hold for 3 seconds and then the subject's head returned passively to neutral position.
  Interventions: Other: Placebo intervention
- Control (No Intervention): The subjects stayed in supine position and no intervention occurred.

INTERVENTIONS:
Other: Cervical spine manual manipulation — In the Manual manipulation group, the thrust was applied in the right side of C3/C4 with neutral flexion/extension, ipsilateral side bending and contralateral rotation. Then, a low amplitude, high velocity thrust in rotation was delivered.
  Arms: Manual manipulation
Other: Cervical spine mechanical manipulation — In the Mechanical manipulation group, the Activator instrument was applied on the right transverse apophyses of C3.
  Arms: Mechanical manipulation
Other: Placebo intervention — The subjects were positioned in the same pre-manipulative position as the manual manipulation group, but the thrust didn't occur. Instead, the position was hold for 3 seconds and then the subject's head returned passively to neutral position.
  Arms: Placebo

SUMMARY:
This study had the goal of analyse the neurophysiologic effects of both mechanical and manual cervical manipulation, in asymptomatic individuals.

DETAILED DESCRIPTION:
In this study, the investigators compared the effects of manual manipulation and instrument assisted manipulation of C3/C4 on muscle tone, elasticity and stiffness and on pressure pain threshold , and pressure pain perception. The muscles evaluated were upper trapezius and biceps brachialis, bilaterally. The study also had a placebo and a control group. All individuals were asymptomatic.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects.
* Minimum of 18 years old.

Exclusion Criteria:

* Pain in cervical region, shoulders or arms.
* History of trauma or disease in the cervical region or upper limb.
* Use of medication that could affect the outcomes (painkillers, NSAID, or anti depressives) during the last week.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2013-05-01 (Actual); Primary Completion 2014-07-01 (Actual); Study Completion 2016-10-01 (Actual)

PRIMARY OUTCOMES:
Pressure pain thresholds | Immediately after the intervention
  To measure the pressure pain threshold, it was used an electronic pressure dynamometer FORCE ONE™ FDIX (Wagner Instruments - Greenwich, USA), with 1cm2 of surface. The values were expressed in Kg/cm2. The pressure was increased at a rate of 1 kg/cm2/s until the subject inform that the sense of pressure has become a sense of pain.
Pressure pain perception | Immediately after the intervention
  To evaluate the pressure pain perception, it was used a Visual Analogue Scale (VAS). The pressure increased until 2,5 kg/cm2 and was hold for 5 seconds, and the subject used the VAS scale to record the pressure pain perception he felt.

SECONDARY OUTCOMES:
Muscle tone | Immediately after the intervention
  To measure muscle tone it was used the MyotonPro device. It was used to evaluate those parameters both on the biceps and on the upper trapezius, bilaterally. The device was located perpendicular to the middle point of each muscle and it were recorded 6 impulses in each one of them. The non-neural tone was recorded as frequency.
Muscle stiffness | Immediately after the intervention
  To measure muscle stiffness it was used the MyotonPro device. It was used to evaluate this parameter both on the biceps and on the upper trapezius, bilaterally. The device was located perpendicular to the middle point of each muscle and it were recorded 6 impulses in each one of them. The muscle stiffness was recorded as N/m.
Muscle elasticity | Immediately after the intervention
  To measure muscle elasticity it was used the MyotonPro device. It was used to evaluate those parameters both on the biceps and on the upper trapezius, bilaterally. The device was located perpendicular to the middle point of each muscle and it were recorded 6 impulses in each one of them. The elasticity was indicated by logarithmic decrement.

CONTACTS AND LOCATIONS:
Overall Officials: Nuno Nogueira, MSc, Principal Investigator — Instituto Politécnico da Saúde do Norte

IPD SHARING:
Plan to Share IPD: No